CLINICAL TRIAL: NCT02212990
Title: Clinical Immunization Safety Assessment (CISA): A Study to Assess the Effect of Prophylactic Antipyretics on Immune Responses and Fever After 2014-2015 and 2015-2016 Inactivated Influenza Vaccine (IIV) Administered to Children 6 Through 47 Months of Age
Brief Title: The Effect of Prophylactic Antipyretics on Immune Responses and Fever After 2014-2015 and 2015-2016 Inactivated Influenza Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00056213; 200-2012-53663 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-04

CONDITIONS: Fever
Keywords: Fever; Antipyretics; Acetaminophen; Ibuprofen; Influenza vaccine; Influenza; Body temperature changes; Signs and symptoms
MeSH Terms: conditions — Fever; Influenza, Human; Body Temperature Changes; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acetaminophen Arm (Active Comparator): Acetaminophen Suspension 160mg / 5mL Oral dose immediately following IIV and every 4 to 6 hours up to 24 hours (Maximum 5 oral doses)
  Interventions: Other: Acetaminophen Arm
- Placebo Arm (Placebo Comparator): Placebo Suspension Oral dose immediately following IIV and every 4 to 6 hours up to 24 hours (Maximum 5 oral doses)
  Interventions: Other: Placebo Arm
- Ibuprofen Arm (Active Comparator): Ibuprofen Suspension 100mg / 5mL Oral dose immediately following IIV and every 6 to 8 hours up to 24 hours (Maximum 4 oral doses)
  Interventions: Other: Ibuprofen Arm

INTERVENTIONS:
Other: Acetaminophen Arm — Blinded Therapy
  Arms: Acetaminophen Arm
Other: Placebo Arm — Blinded Therapy
  Arms: Placebo Arm
Other: Ibuprofen Arm — Open Label Therapy
  Arms: Ibuprofen Arm

SUMMARY:
This study aims to conduct a double-blind, placebo-controlled study to assess the effect of prophylactic antipyretics on the immune responses and rates of fever after inactivated influenza vaccine (IIV) in children 6 through 47 months of age.

In this study, 160 healthy children, 6 through 47 months of age, including some children at risk of febrile seizure, will be randomized to one of three different treatment arms. Children will receive either blinded therapy with prophylactic acetaminophen or placebo immediately following and every 4 to 6 hours in the 24 hours after receipt of a dose of IIV or open-label ibuprofen every 6 to 8 hours in the 24 hours after receipt of a dose of IIV. Children will be followed for the occurrence of fever, fussiness, changes in appetite and sleep patterns, and use of medical services on the day of and for two days following vaccination. Antibody to influenza antigens contained in the respective 2014-2015 and 2015-2016 vaccines as measured by hemagglutination inhibition (HAI) antibody will be assessed at baseline and four weeks following vaccination. The proportions of children experiencing fever, having solicited side effects, using medical services, demonstrating a serologic response corresponding to seroprotection and seroconversion to each of the IIV antigens will be determined for groups of children in each of the three treatment arms. Likewise geometric mean HAI titers (GMTs) and corresponding 95% confidence intervals for each IIV antigen will be calculated for the three treatment arms. The investigators hope to learn whether or not prophylactic antipyretics affect the immune response and fever rates following IIV.

ELIGIBILITY:
Inclusion Criteria:

1. The child must be 6 through 47 months of age.
2. The child must weigh 5.4 kilograms.
3. The child must be receiving IIV this season.
4. If the child is two years of age or older and needs two doses of influenza vaccine this season the parent/guardian intends for the child to receive IIV for the second dose.
5. The parent/guardian must be willing and capable of providing written informed consent for the child.
6. The parent/guardian must be available for follow-up and must at minimum have telephone access.
7. The parent/guardian must agree to sign a medical release for the child so that study personnel may obtain medical information about the child's health (if needed).

Exclusion Criteria:

1. History of receipt of current year's licensed influenza vaccine.
2. Planned receipt of the live attenuated nasally administered influenza vaccine this year
3. History of a severe allergic reaction (e.g. anaphylaxis) to any component of influenza vaccine, including egg protein, formaldehyde, octylphenol ethoxylate, gelatin, or thimerosal if using thimerosal containing vaccine.
4. History of a severe allergic reaction (e.g. anaphylaxis) following a prior dose of influenza vaccine.
5. History of an allergic reaction following acetaminophen or ingredients in the acetaminophen product.
6. History of an allergic reaction following ibuprofen or ingredients in the ibuprofen product.
7. History of an allergic reaction following aspirin or other pain reliever or fever reducer.
8. History of liver disease.
9. Currently taking the blood thinning drug warfarin (Coumadin) or other blood thinners.
10. History of recent or planned heart surgery within the past 3 months or next 3 months.
11. History of stomach ulcer or bleeding problem.
12. Currently already routinely taking prescription or nonprescription non-steroidal anti-inflammatory drugs or NSAIDs (aspirin, ibuprofen, naproxen, or others)
13. Received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination in this study or expects to receive a licensed vaccine during the 28 days following the last influenza vaccination in this study. Concomitant vaccinations are not allowed.
14. Routine immunizations are delayed or will be delayed by not being able to receive a concomitantly administered vaccine or a needed vaccine in the 28 days following the last influenza vaccination in this study.
15. Received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to vaccination in this study, or expects to receive an experimental/investigational agent within the follow-up time period (28 days after the last vaccination in this study).
16. A moderate to severe acute illness and/or a reported temperature greater than or equal to 100.0°F (37.8°C) within 72 hours prior to first dose of IIV or an axillary temperature greater than or equal to 100.0°F (37.8°C) at the time of enrollment. (This may result in a temporary delay of vaccination. For those needing a second dose of IIV, a moderate to severe acute illness and/or a reported temperature greater than or equal to 100.0°F (37.8°C) within 72 hours prior to second dose of IIV may result in a temporary delay of vaccination).
17. Receipt of an antipyretic medication (acetaminophen or ibuprofen) within 72 hours prior to the first dose of IIV (This may result in a temporary delay of vaccination) or is already planning to administer a prophylactic antipyretic medication on the day of and the day following any dose of IIV (this exclusion does not apply if the caretaker indicates he/she might administer antipyretics after vaccination to reduce a fever).
18. Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
19. Long term (at least 14 days of prednisone 2 mg/kg/day or equivalent other glucocorticoid), any parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (topical and nasal steroids are allowed).
20. History of Guillain-Barré syndrome within 6 weeks of a prior dose of influenza vaccine.
21. Has any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Seroconversion | One month following the last dose of IIV
  Seroconversion (an HAI titer ≥ 1:40 four weeks post- vaccination if the baseline titer is < 1:10 or a four-fold rise in HAI titer if the baseline titer is ≥ 1:10) for each IIV antigen

SECONDARY OUTCOMES:
Seroprotection | One month following the last dose of IIV
  Seroprotection (the proportion of subjects with an HAI titer >1:40) to each IIV antigen
Geometric mean HAI titer | One month following the last dose of IIV
  Geometric mean HAI titer (GMT) and 95% confidence interval for each IIV antigen

OTHER OUTCOMES:
Fever | Days 0, 1, and 2 following IIV
  Proportions of children with fever (≥ 38°C and ≥ 39°C) on days 0, 1, and 2 following IIV
Systemic symptoms following IIV | Days 0, 1, and 2 following IIV
  Proportions of children with fussiness, appetite change, or altered sleep on days 0, 1, and 2 following IIV
Receipt of medical attention | Days 0, 1, and 2 following IIV
  Proportions of children receiving medical attention on days 0, 1, and 2 following IIV

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, MPH, Principal Investigator — Duke Unviersity School of Medicine; Karen Broder, MD, Principal Investigator — Centers for Diseaes Control and Prevention
Locations (1):
- Duke University Health System, Durham, North Carolina, United States